CLINICAL TRIAL: NCT00974714
Title: Effects of Oral L-arginine on Chronic Hypertension in Pregnancy
Brief Title: L-arginine Effects on Chronic Hypertension in Pregnancy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Facchinetti Fabio, University of Modena and Reggio Emilia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Facchinetti; Neri Isabella (Other Grant/Funding Number: Fabio Facchinetti); De Pace Viviana (Other Grant/Funding Number: Fabio Facchinetti); Monari Francesca (Other Grant/Funding Number: Fabio Facchinetti); Dante Giulia (Other Grant/Funding Number: Fabio Facchinetti)
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2009-09

CONDITIONS: Hypertension in Pregnancy
Keywords: chronic hypertension in pregnancy
MeSH Terms: conditions — Hypertension, Pregnancy-Induced | interventions — Arginine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Oral L-arginine 2 g twice a day, for 14 weeks
  Interventions: Drug: L-arginine
- 2 (Placebo Comparator): oral placebo twice a day for 14 weeks
  Interventions: Other: placebo

INTERVENTIONS:
Drug: L-arginine — Oral L-arginine 2 g twice a day for 14 weeks
  Arms: 1
Other: placebo — oral placebo 2 g twice a day for 14 weeks
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the effects of oral L-arginine administration on pregnant women at second trimester of gestation with chronic hypertension, respect with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between 18-20 weeks of gestation with chronic hypertension

Exclusion Criteria:

* Other maternal or fetal systemic disease

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-09; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
to evaluate blood pressure changes during oral L-arginine or placebo administration in pregnant women with chronic hypertension at second trimester of gestation | 14 weeks

SECONDARY OUTCOMES:
evaluate if is necessary to add a conventional therapy for hypertension, to evaluate pregnancy outcomes and eventual complications, to evaluate safety of oral L-arginine administration | 14 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - University of Modena and Reggio Emilia, Modena, Emilia-Romagna
  - University of Modena and Reggio Emilia, Modena, Mo